CLINICAL TRIAL: NCT04577534
Title: COVID-19: Salvage TOcilizumab as a Rescue Measure. Use of Tocilizumab in the Inflammatory Phase of COVID-19 / New Coronavirus Disease
Brief Title: COVID-19: Salvage TOcilizumab as a Rescue Measure
Acronym: COVIDSTORM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jarmo Oksi (Other Government)
Responsible Party: Sponsor-Investigator, Jarmo Oksi, Head of Infectious Diseases, Turku University Hospital
Organization: Turku University Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2020-002039-31; 2020-002039-31 (EudraCT Number); T124/2020 (Other: Turku University Hospital); KLnro 36/2020 (Other: Fimea); dnro 68/06.00.01/2020 (Other: TUKIJA / VALVIRA)
Record Dates: First submitted 2020-09-03; First posted 2020-10-08 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: COVID-19; new coronavirus disease; tocilizumab
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab (TCZ) (Experimental): Participants will receive one infusion of iv TCZ (according to weight of patient)
  Interventions: Drug: iv Tocillizumab (TCZ)
- standard of care (no TCZ) (No Intervention): Participants will receive standard of care

INTERVENTIONS:
Drug: iv Tocillizumab (TCZ) — Participants are randomized (2:1) to receive TCZ or Standard of Care
  Arms: Tocilizumab (TCZ)

SUMMARY:
Evaluating the efficacy of Tocilizumab in hospitalized patients in the inflammatory phase of COVID-19. Randomization 2:1 (TCZ:standard of care).

ELIGIBILITY:
Inclusion Criteria:

* written informed consaent obtained
* hospitalized with COVID-19 disease
* Age >/= 18 years
* SARS CoV-2 NhO posit
* Sp=2 </93% on ambient air or respiratory rate >30 /min
* Any 2 of the 4: P-IL-6 > 2 x ULN / P-ferritin > 2 x ULN / P-FIDD >1.5 mg/l / P- CRP >40 mg/l without obvious presence of bacterial infection (normal values: P -IL-6 <5.9 ng/l; P-ferritin, men 30-400 mikrog/l, women 13-150 mikrog/l ; P-FIDD (Fibrin degradation products, D-dimer) <0.5 mg/l; P-CRP <10 mg/l)

Exclusion Criteria:

* Known severe allergic reactions to monoclonal antibodies
* Active confirmed tuberculosis with ongoing treatment or obvious tuberculosis or obvious other bacterial, fungal or viral infection (besides COVID-19)
* In the opinion of the clinical team, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Long-term oral anti-rejection or immunomodulatory drugs (including corticosteroids equivalent to methylprednison 15mg/day)
* Pregnant or lactating women. If needed, exclusion of pregnancy should be performed by laboratory test (U-hCG-O).
* Participating in other drug clinical trials
* Absolute neutrophil count < 1 x10E9/l
* Platelet count <50 x10E9/l
* ALAT >10x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Clinical status at day 28 | day 28
  (assessed using 7-category ordinal scale) 7 death 6 in ICU with ECMO/ mechanical ventilation 5 in ICU, no ECMO/ mechanical ventilation 4 in hospital, not ICU, needs supplementary oxygen 3 in hospital, not ICU, no supplementary oxygen 2 not in hospital, but not back to normal
  1 not in hospital, back to normal

SECONDARY OUTCOMES:
Time to clinical improvement | 28 days
  defined as a National Early Warning Score 2 (NEWS2) of>/=2 maintained for 24 hours
Time to decline of at least 2 categories | 28 days
  relative on a 7-category ordinalscale of clinical status
Incidence of mechanical and/or non-invasive ventilation | 28 days
  (mode and duration of respiratory support) Hospital day when respiratory support needed with non-invasive ventilation - and duration.
  Hospital day when respiratory support needed by invasive mechanical ventilation -and duration.
Number of ventilator-free days to day 28 | 28 days
  days not in ventilator
Organ failure free days to day 28 | 28 days
  days without organ failure
Incidence of ICU stay | 28 days
  ICU admission day
Duration of ICU stay | 28 days
  days on ICU
Time to clinical failure | 28 days
  time to death, mechanical ventilation, or ICU admission (whichever occurs first)
SAPS II | 28 days
  during ICU stay SAPS II = simplified acute physiology score II min 0 (best), max 163 (worst)
CCI | 28 days
  during ICU stay CCI = Charlson Comorbidity Index min 0 (best), max 37 (worst)
APACHE II | 28 days
  during ICU stay APACHE II = acute physiology and chronic health evaluation II min 0 (best), max 71 (worst)
SOFA 6 | 28 days
  during ICU stay SOFA 6 = sequential organ failure assessment min 0 (best), max 24 (worst)
Mortality rate | 28 days
  during and end of period of 28 days
Time to hospital discharge or "ready for discharge" | 28 days
  as evidenced by normal body temperature and respiratory rate and stable oxygen saturation on ambient air or </=2 l supplemental oxygen
Duration of supplemental oxygen | 28 days
  days on suppl oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided
plan to investigate if it is possible by law